CLINICAL TRIAL: NCT00772798
Title: A Phase I/II Non-Comparative Study of Paclitaxel Plus Carboplatin in Combination With Vorinostat in Patient With Advanced, Recurrent, Epithelial Ovarian Cancer
Brief Title: A Phase I/II Study of Paclitaxel Plus Carboplatin Plus Vorinostat in Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Jørn Herrstedt, M.D., DMSCI, professor, dept. of oncology, Odense University Hospital, Sdr. Boulevard 29, DK-5000 C, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S9X
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; HDAC inhibitor; vorinostat
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Carboplatin; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Paclitaxel, Carboplatin and Vorinostat — Intravenous paclitaxel (175 mg/m2) and carboplatin (AUC 5) and oral vorinostat 400 mg day 1-14 every three weeks.
  Other Names: Taxol; Carboplatin; Vorinostat

SUMMARY:
TITLE:A Phase II non-comparative study of paclitaxel plus carboplatin in combination with Vorinostat in patients with advanced, recurrent epithelial ovarian cancer. INDICATION:Second-line treatment of patients with recurrent platinum-sensitive epithelial ovarian cancer. RATIONALE:Recurrent epithelial ovarian cancer is today an incurable disease. The current standard of care consists of systemic chemotherapy using either carboplatin plus paclitaxel (in platinum-sensitive patients) or single agent chemotherapy with agents like liposomal doxorubicin, topotecan, weekly paclitaxel or gemcitabine (platinum non-sensitive patients). The outcome for patients with advanced ovarian cancer nevertheless remains poor.Preclinical evidence suggests that vorinostat, a potent histone deacetylase (HDAC) inhibitor, may potentiate the antitumor activity of paclitaxel and/or carboplatin. The study will assess whether the addition of vorinostat to paclitaxel plus carboplatin is manageable and induces reasonable response rates in patients with advanced recurrent, platinum-sensitive ovarian cancer. Biomarkers will be collected from both primary tumors and biopsies before and after start of treatment with vorinostat.

DESIGN:Phase II, single-center study. All eligible patients will be treated with intravenous paclitaxel plus carboplatin plus oral vorinostat. Patients will be treated with a maximum of 6 cycles or until disease progression, unacceptable toxicity or withdrawal of consent. Clinical endpoints will include adverse experiences, progression-free survival (PFS) and response rate (RR). SAMPLE:Patients must have a histologically confirmed diagnosis of epithelial ovarian cancer, cancer of the Fallopian tube or primary peritoneal adenocarcinoma. All patients will have received first-line therapy with carboplatin plus paclitaxel. Patients should be platinum sensitive, defined as recurrence or progression of ovarian cancer, cancer of the Fallopian tubes or primary peritoneal adenocarcinoma 6 months or later after the end of first-line chemotherapy. Patients to be enrolled on this study must have acceptable performance status and acceptable renal and hepatic function, and be free of other serious intercurrent illness that could impair their ability to receive protocol therapy. The study will include up to 55 assessable patients, of which 20 will provide biomarkers. It is estimated that the inclusion period will last approximately 24 months. DOSAGE/DOSAGE FORM, ROUTE, AND DOSE REGIMEN Eligible patients will be treated with paclitaxel (175 mg/m2) and carboplatin AUC5 administered by intravenous infusion (IV) on day 1 of each treatment cycle. In addition, all eligible patients will receive treatment with oral vorinostat (400 mg) administered once daily by mouth with food on days -4 through 10 of Cycle 1 (25-day treatment cycle) and days 1 through 14 of each subsequent 21-day treatment cycle. Patients will receive antiemetic therapy according to institutional guidelines as well as premedication with dexamethasone, and antihistamines (an H1-receptor antagonist and an H2-receptor antagonist) for prevention of the side effects of paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Histological verified epithelial carcinoma derived from ovarian, peritoneum or uterine tubes
2. Women ≥18 years old.
3. ECOG performance status ≤2.
4. Expected duration of life >3 months.
5. Previous treatment regimen containing platinum and paclitaxel.
6. Platinum and paclitaxel sensitive tumor, defined as a minimum of 6 months from cessation of treatment until disease progression.
7. Measurable or assessable lesion.Patients having increased CA-125 as the only sign of recurrence are also eligible.
8. Normal organ functions defined by the following values:

   Absolute neutrophil count (ANC) ≥1,500/µL Platelets ≥100,000/µL Hemoglobin ≥9.0g/dL or > 5.7 mmol/L CA125 0-35 Glomerular filtration rate (GFR) measured using Cr-EDTA clearance GFR ≥50 mL/minute (not corrected for body surface area) Serum Total bilirubin ≤1.5 times the ULN AST (SGOT) and ALT (SGPT) ≤2.5 times the ULN Alkaline phosphatase ≤5.0 times the ULN Prothrombin time (PT) ≤1.2 times the ULN unless the patient is receiving therapeutic anticoagulation.

   Partial thromboplastin time (PTT) ≤1.2 times the ULN unless the patient is receiving therapeutic anticoagulation.
9. Signed informed consent before inclusion.
10. Prepared to appear for the planned follow-up visits and capable of handling toxicity.

Exclusion Criteria:

1. Patients treated with an experimental drug within the last 4 weeks before inclusion, and patients who receive other concomitant anticancer treatment.
2. Patients having an active infection, or who have received intravenous antibacterial or antifungal medicine within the last 2 weeks before inclusion.
3. Patients previously treated with an HDAC inhibitor. Patients, who have been treated with Valproate for convulsions can be included, however only if the treatment has taken place > 30 days before inclusion.
4. Patients treated with steroid, who are not stabilized on a firm dose equivalent to a maximum of 10 mg prednisolone per day for the last 4 weeks before inclusion.
5. Previous treatment with more than first-line chemotherapy.
6. Progression during treatment with first-line chemotherapy containing platin/paclitaxel or disease progression less than 6 months after treatment cessation.
7. Concomitant serious and/or non-controllable medical condition such as non-controllable infection (including HIV infected patients), hypertension, ischemic heart disease, myocardial infarction within the last 6 months, congestive heart failure.
8. Previous treatment for, or other concomitant malignant disease within the last 5 years, except for curative treated carcinoma in situ cervical cancer or basal cell carcinoma.
9. Previous severe allergic reactions in connection with carboplatin, paclitaxel or agents within the histone deacetylase inhibitor group.
10. Women of child-bearing age. Women must have undergone surgical removal of the ovaries or be post-menopausal with no menstruation during the previous year.
11. Peripheral neuropathy ≥ grade 2, unless this is due to a medical condition.
12. Patients with history of severe hyper sensitive reactions with regards to products containing Cremophor EL (cyclosporine or K-vitamin) and/or patients with known hypersensitivity towards agents chemically connected to paclitaxel, carboplatin or vorinostat.
13. Patients with known cerebral metastases or clinical signs of cerebral metastases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Primary: To assess the objective response rate, safety, tolerability, and adverse experience profile of vorinostat administered in combination with paclitaxel plus carboplatin in patients with platin sensitive recurrent epithelial ovarian cancer. | Until disease progression

SECONDARY OUTCOMES:
To determine the progression-free survival (PFS) of patients with advanced, recurrent epithelial ovarian cancer, cancer of the Fallopian tube or primary peritoneal adenocarcinoma treated with paclitaxel plus carboplatin and vorinostat. | Until progression of disease

CONTACTS AND LOCATIONS:
Overall Officials: Jørn Herrstedt, professor, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Oncology R, Odense, Denmark